CLINICAL TRIAL: NCT01421433
Title: Non Inferiority,Phase III,Multicentric,Double Blind,Randomized,Parallel Study,Comparing Dolamin Flex (Lysine Clonixinate+Cyclobenzaprine) and Tandrilax(Caffeine +Carisoprodol+Diclofenac+Paracetamol)in Pain Reduction in Patients With Lumbago
Brief Title: A Comparative Study Between Lysine Clonixinate+Cyclobenzaprine and Caffeine+Carisoprodol+Sodium Diclofenac+Paracetamol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Farmoquimica S.A. (Industry)
Collaborators: Pharmagenix Projetos em Medicina Farmacêutica Ltda. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FQM 01/11
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Low Back Pain
Keywords: Clonixin; Anti-Inflammatory Agents, Non-Steroidal; Cyclooxygenase Inhibitors; Lysine; L-Lysine; Lysine Acetate; Lysine Hydrochloride; Amitriptyline
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tandrilax (Active Comparator): Reference product Intervention: Drug: Tandrilax (caffeine+carisoprodol+sodium diclofenac+paracetamol)
  Interventions: Drug: Tandrilax
- Dolamin Flex (Experimental): Test product Intervention: Drug: Dolamin Flex (Lysine clonixinate and cyclobenzaprine)
  Interventions: Drug: Dolamin Flex

INTERVENTIONS:
Drug: Tandrilax — Tandrilax (caffeine, carisoprodol, sodium diclofenac, paracetamol). Tablets, administered 3 times a day, for 7 consecutive days.
  Arms: Tandrilax
Drug: Dolamin Flex — Dolamin Flex (lysine clonixinate and cyclobenzaprine). Tablets, administered 3 times a day, for 7 consecutive days.
  Arms: Dolamin Flex

SUMMARY:
Non inferiority, multicentric, double blind study whose the primary objective is to compare the effectiveness of two products in pain reduction. Primary endpoint: reduction in pain average at day 7 compared to day 1(baseline), using Analogue Visual Scale (AVS) for pain evaluation. Secondary endpoint: to evaluate the products safety at the gastrointestinal system.

DETAILED DESCRIPTION:
Phase IIIb, non-inferiority, multicentric, double-blind study.Population: 160 patients, 80 in each study arm, both gender with mild to moderate lumbago, without irradiation and with muscle contraction, aged 18 (eighteen) and 65 (sixty five) years, without previous history of stomach or duodenal ulcer and gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the nature of the study and given written informed consent
* Patients with mild to moderate lumbago
* Aged between 18 and 65 years old

Exclusion Criteria:

* Known allergy or sensitivity to drug components
* Treatment with another anti inflammatory or corticoid
* Treatment with oral anticoagulants
* Treatment with oxidase monoamine 2 weeks before the study
* Treatment with methotrexate
* Stomach or duodenal ulcer and gastritis
* Dehydration
* Acute myocardial infarction or heart failure
* Hyperthyroidism
* Pregnant or lactating patients
* Treatment with lithium
* User of alcohol and barbiturates
* Hepatic or renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-08 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pain average reduction | 7 days
  The metric that will be used is Pain Analog Visual Scale (PAVS), that it is a graphical representation with values 0-10.
  To use the PAVS, the principal investigator should question the patient regarding their pain level, and the value 0 (zero) means no pain and the value 10 (ten) indicates the maximum pain level.

SECONDARY OUTCOMES:
Identification of possible gastrointestinal effects | 7 days
  The metric that will be used is checking the safety data reported by the patient in the Patient Diary and / or using data reported by patients by Phone Call.
  A diary will be given for the patient, to make notes about possible gastrointestinal adverse events.
  The principal investigator should call to the patient to know about possible gastrointestinal adverse effects of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio T. Silva, Phd, Principal Investigator — Hospital São Luiz
Locations (1):
- Hospital São Luiz, São Paulo, São Paulo, Brazil